CLINICAL TRIAL: NCT06620796
Title: A Phase II Study of Ivonescimab Combined with Cadonilimab and Chemotherapy in Extensive-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of the Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024LY0857
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: SCLC, Extensive Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1 (Experimental): Ivonescimab (20 mg/kg, IV, every 3 weeks) plus platinum-based chemotherapy (carboplatin [area under the curve (AUC) 5 mg/mL per min, IV] and etoposide [100 mg/m2, IV, D1-D3] for ES-SCLC) for up to four cycles, followed by maintenance therapy with cadonilimab (10 mg/kg, IV, every 6 weeks, D2) and Ivonescimab (20 mg/kg, IV, every 3 weeks, D1) .
  Interventions: Drug: Arm 1
- Arm2 (Experimental): Cadonilimab (10 mg/kg, IV, every 6 weeks, D2) and Ivonescimab (20 mg/kg, IV, every 3 weeks, D1) plus paclitaxel [260 mg/m2, IV, D1].
  Interventions: Drug: second-line group

INTERVENTIONS:
Drug: Arm 1 — Ivonescimab combined with Cadonilimab plus EC
  Other Names: AK112+AK104 group
  Arms: Arm1
Drug: second-line group — AK112+AK104+paclitaxel
  Other Names: AK112+AK104+paclitaxel
  Arms: Arm2

SUMMARY:
The goal of this clinical trial is to investigate the efficacy, safety and tolerability of Ivonescimab combined with Cadonilimab and chemotherapy in extensive-stage small cell lung cancer patients. And also explore the potential biomarkers for predicting the efficacy of Ivonescimab combined with Cadonilimab for extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before implementing any trial-related procedures;
* Aged 18-80 years;
* Expected survival of more than 3 months;
* histologically or cytologically confirmed ES-SCLC according to the American Veterans Cancer Association VALG staging system；
* Arm 1: subjects who have not received previous systemic therapy for extensive-stage SCLC; Or patients who had received definitive chemoradiotherapy for limited-stage small cell lung cancer but had disease progression > 6 months later;Arm 2：ES-SCLC patients who progressed after only one PD-1/PD-L1 combination chemotherapy and had response to previous treatment (PFS ≥ 3 months), no more than two systemic chemotherapy regimens were used；
* The investigator confirms the presence of at least one measurable lesion according to RECIST 1.1 criteria;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Adequate hematologic function, defined as absolute neutrophil count (ANC) >= 1.5 x 10^9/L, platelet count >= 100 x 10^9/L, hemoglobin >= 90 g/L (without transfusion history within 7 days);
* Adequate liver function, defined as total bilirubin level <= 1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels <= 2.5 times ULN in all patients, or <= 5 times ULN in patients with liver metastases;
* Adequate renal function, defined as serum creatinine <= 1.5 times ULN;
* Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) <= 1.5 times ULN; for subjects receiving anticoagulant therapy, INR/PT should be within the range planned by the anticoagulant;
* Women of childbearing potential must have a negative pregnancy test within 7 days before starting treatment, and must use reliable contraceptive measures (such as intrauterine device, contraceptive pills, and condoms) during the trial and for 30 days after the end of the trial; male subjects of reproductive potential must use condoms for contraception during the trial and for 30 days after the end of the trial;
* Willingness to comply with regular follow-up visits and trial requirements.
* Participants were required to provide 10 or more unstained FFPE pathological slides (preferably newly obtained tumor tissue) archived or freshly obtained within 3 months prior to the first dose of medication. Tumor lesions used for fresh-tissue biopsy should not be used as RECIST v1.1 target lesions unless they are the only measurable lesion. The collection of archived tumor-tissue samples beyond 3 months of age was permitted, with the consent of the medical monitor, if no samples were available within 3 months of age and biopsy, as judged by the investigator, might increase the risk to the subject. If more than 10 slides were not available, some or all of the slides could be waived with investigator approval；
* Participants were required to provide approximately 10 unstained FFPE tumor tissue slides for efficacy biomarker exploration. If it cannot be provided, it can be exempted after approval from the investigator and will not affect the Participants participation in this study；

Exclusion Criteria:

* Currently participating in interventional clinical research treatment;
* For Arm 1: a) Prior immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1 /L1 antibody, anti-CTLA-4 antibody, anti-TIGIT antibody, anti-LAG-3 antibody, etc.), immune checkpoint agonists (e.g. ICOS, CD40, CD137, GITR, OX40 antibody, etc.), immune cell therapy, and any treatment targeting the tumor immune mechanism; b) previous systemic anti-angiogenic therapy, including but not limited to bevacizumab small molecule TKI, etc. For Arm 2:

  a) PD-1/L1 inhibitor crossover therapy: after the failure of PD-1/L1 inhibitor combined with chemotherapy, the chemotherapy regimen was changed and the original PD-1/L1 inhibitor was given again. b) Prior immunotherapy other than PD-1/L1 inhibitors, including immune checkpoint inhibitors (e.g., anti-TIGIT antibody, anti-LAG-3 antibody, etc., anti-CTLA-4 monoclonal antibody), immune checkpoint agonists (e.g. ICOS, CD40, CD137, GITR, OX40 antibody, etc.), immune cell therapy, and any treatment targeting the mechanism of tumor immune action. c) previous treatment with a taxol chemotherapeutic agent. d) previous systemic anti-angiogenic therapy, including but not limited to bevacizumab, small molecule TKI, etc.
* Imaging during the screening period showed that the tumor was surrounded by important blood vessels or had obvious necrosis or cavities, and the investigator judged that the entry of the study would cause bleeding risk.
* active autoimmune disease requiring systemic treatment within the past 2 years (e.g., with disease-modifying medications, corticosteroids, immunosuppressants). Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) is not considered a systemic treatment.
* history of noninfectious pneumonia/interstitial lung disease requiring systemic glucocorticoid treatment or current noninfectious pneumonia.
* History of brain stem, meningeal metastasis, spinal cord metastasis or compression.presence of active central nervous system (CNS) metastases; Participants who had previously been treated for brain metastases (e.g., surgery, radiotherapy) were allowed if they were clinically stable for at least two weeks after treatment (calculated from the time of the first administration of the study drug) and if corticosteroids were discontinued 7 days before the administration of the study drug. Participants with untreated, asymptomatic brain metastases (i.e., no neurologic symptoms, no need for corticosteroids, no brain metastases measuring >1.5 cm in the greatest dimension, and no substantial premetastatic edema) were eligible for enrollment
* presence of current uncontrolled coexisting medical conditions, including but not limited to decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorder, severe active peptic ulcer disease, or gastritis, or mental illness/social condition that would limit compliance with study requirements or affect the participant's ability to provide written informed consent;
* previous history of myocarditis, cardiomyopathy, and malignant arrhythmia. The presence of unstable angina, myocardial infarction, congestive heart failure (New York Heart Association functional class 2 or higher), or vascular disease (e.g., aortic aneurysm at risk for rupture) that required hospitalization within 12 months before the first dose of the study drug or other cardiac impairment (e.g., uncontrolled arrhythmias, myocardial ischemia) that could affect the safety evaluation of the study drug; The patient had a history of esophagogastric varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months before the first dose of medication. Any arterial thromboembolic event, venous thromboembolic event of NCI CTCAE version 5.0 or higher, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy occurred 6 months before the first dose. An acute exacerbation of chronic obstructive pulmonary disease occurred within 1 month before the first dose, except for infusion-related thrombosis that had occurred for more than 4 weeks.
* history of severe bleeding tendency or coagulopathy; Clinically significant bleeding symptoms within 1 month before the first dose of medication, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or coughing up ≥1 teaspoon of blood or small blood clot or only coughing up blood without sputum, and those with blood in sputum were allowed), nasal bleeding (excluding epistaxis and retraction of nasal bleeding); Continuous antiplatelet or anticoagulant therapy had been administered within 10 days before the first dose.
* lack of resolution of toxicity from prior antineoplastic therapy, defined as failure to return to NCI CTCAE version 5.0 grade 0 or 1 or levels specified in the inclusion/exclusion criteria, with the exception of alopecia. Subjects with irreversible toxicity that was not expected to worsen with study drug administration (e.g., hearing loss) may be enrolled after consultation with the medical monitor. Subjects with long-term radiation-induced toxicity that, in the judgment of the investigator, did not recover from, may be included in the study.
* serious infection within 4 weeks before the first dose, including but not limited to coexisting conditions requiring hospitalization, sepsis, or severe pneumonia; Active infection (excluding antiviral therapy for hepatitis B or hepatitis C) that had received systemic anti-infective therapy within 2 weeks before the first dose.
* history of immunodeficiency; HIV antibody positive; Long-term use of systemic corticosteroids or other immunosuppressive agents is ongoing.
* Subjects with known active pulmonary tuberculosis should be excluded by clinical examination (e.g., sputum test, chest X-ray, etc.); Known active syphilis infection.
* history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* presence of pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage.
* subjects with active hepatitis B (HBsag-positive and HBV-DNA > 500 copies /ml or higher than the lower limit of detection); Subjects with active hepatitis C (HCV antibody-positive).
* had a major surgical procedure or major trauma within 30 days before or within 30 days after the first dose (at the discretion of the investigator); Minor local procedures (excluding peripherally inserted central catheters and intravenous-access ports) had been performed within 3 days before the first dose.
* received live attenuated influenza vaccine within 30 days before the first dose or plan to receive live attenuated influenza vaccine during the study and cannot receive live attenuated influenza vaccine within 90 days after treatment after the last dose of the study drug.
* known allergy to any component of any study drug; A history of severe hypersensitivity reactions to other monoclonal antibodies was known.
* known history of mental illness, substance abuse, alcohol or drug abuse.
* pregnant or lactating women.
* The presence of any past or current medical conditions, treatments, or laboratory abnormalities that may confound the results of the study, preclude full participation in the study, or participation in the study may not be in the best interest of the subject

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
6-month Progression-Free Survival (PFS) rate | 6-month
  The 6-month Progression-Free Survival (PFS) rate refers to the proportion of patients who are alive and without disease progression six months after starting treatment.

SECONDARY OUTCOMES:
Progression-free Survival | up to 60 months
  Progression-free survival measures the length of time during and after treatment that a patient lives with the disease without it progressing.
objective response rate | up to 24 months
  Objective response rate represents the proportion of patients showing a predefined level of tumor shrinkage or disappearance in response to treatment.
Overall Survival | up to 100 months
  Overall survival measures the length of time from the start of treatment until death from any cause, indicating the effectiveness of the treatment in prolonging patients' lives.
duration of response | up to 24 months
  Duration of response refers to the length of time during which a patient's tumor remains in remission or shows a positive response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxia Su, Doctor, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Public article
Supporting Information: Study Protocol
Time Frame: 2025.9-2027.9
Access Criteria: send request to research team for access to the data